CLINICAL TRIAL: NCT05528874
Title: Glycemic Index Analysis of Functional Bakery Products on a Group of Healthy Volunteers, a NUTRACORE Study
Brief Title: NUTRACORE, Glycaemic Index and Appetite
Acronym: NTRCR-vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Polo AgriFood - Miac Scpa (Unknown); Albertengo Panettoni (Unknown)
Responsible Party: Principal Investigator, Flavia Prodam, Associated Prof. in Clinical Nutrition and MD, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CE 054/2022
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hyperglycemia; Hyperglycemia, Postprandial; Appetitive Behavior; Hyperinsulinism; Consumer Preference
MeSH Terms: conditions — Hyperglycemia; Appetitive Behavior; Hyperinsulinism; Consumer Behavior

STUDY DESIGN:
Intervention Model Description: This study is composed by 2 parts. The same participants are enrolled in a single arm study (5 days), followed by a cross-over part (2 days)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subject and investigators cannot know which of the last 2 formulations are given and the unmasking will be made by the coordinator group of Nutracore project
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: randomized to receive recipe 4 after the 5 days single arm study, and then recipe 5 (Experimental): Healthy volunteers that signed informed consent. Will consume all recipes in crescent order.
  Interventions: Dietary Supplement: Same intervention for both groups: glycaemic index assessment of 3 biscuits recipes; Dietary Supplement: Crossover: Recipe 4 before recipe 5
- Group 2: randomized to receive recipe 5 after the 5 days single arm study, and then recipe 4 (Experimental): Same as before but randomized to receive recipe 5 before recipe 4.
  Interventions: Dietary Supplement: Same intervention for both groups: glycaemic index assessment of 3 biscuits recipes; Dietary Supplement: Crossover: Recipe 5 before recipe 4

INTERVENTIONS:
Dietary Supplement: Same intervention for both groups: glycaemic index assessment of 3 biscuits recipes — Following International standards ISO 26642 guidelines, subjects (at fasting) will have their glycemia measured and after will consume a solution containing 50g of glucose and 100g of water. In the following 2 hours, glycemia and other blood parameters will be taken 6 times (at 15, 30, 45, 60, 90, and 120 minutes). This protocol is repeated twice within 3 months. After these 2 days, with the same methods, they will come to our clinic to test 3 different recipes of biscuits (characteristics are presented on request). Subjects and investigators are not blinded to these biscuits characteristics.
  Other Names: Recipe 1,2,3
Dietary Supplement: Crossover: Recipe 4 before recipe 5 — After the assessment of fasting parameters, subjects will consume recipe 4 (chocolate biscuits) and perform a 180 min curve with blood taken at 15, 30, 45, 60, 90, 120, and 180 minutes. In this case, both investigators and patients are blinded to the presence of an additional "non-nutritive, non-toxic and without taste" encapsulated bitter compound (artemisia absinthium), that could be present in recipe 4 or recipe 5. On the second day (with at least a week gap), patients will consume recipe 5. Questionnaires and a food diary will also be requested for subjects for lunch and dinner.
  Other Names: Recipe 4-5
  Arms: Group 1: randomized to receive recipe 4 after the 5 days single arm study, and then recipe 5
Dietary Supplement: Crossover: Recipe 5 before recipe 4 — Same as previous group, but starting with recipe 5
  Other Names: Recipe 5-4
  Arms: Group 2: randomized to receive recipe 5 after the 5 days single arm study, and then recipe 4

SUMMARY:
In recent decades, the world prevalence of obesity and type 2 diabetes (DMT2) has increased dramatically, resulting in a global epidemic. One of the aspects more connected to the etiology of these pathologies is undoubtedly the concept of the glycemic index (GI) and glycemic load (CG). It has been shown that, with the same CG, that is of carbohydrates contained in a food, a food with a higher GI tends to raise blood sugar more quickly (and consequently insulin), causing several negative effects on the body. We now have sufficient evidence to show that high GI diets are associated with increased incidence of DMT2, hyperlipoproteinemia, and cardiovascular disease.

Although simple carbohydrates, namely sugars, have always been considered the major inducers of hyperglycemia and hyperinsulinemia, in reality also starches, or complex carbohydrates digestible by humans, may lead to an increase in blood sugar levels which is not as rapid but often equally harmful to health, since the GC is generally higher.

The reason why a high GI diet is responsible for this increased risk of developing pathologies is not unambiguous. We can identify at least 4 probable mechanisms.

1. Sudden hyperglycemia tends to cause insulin to rise beyond what is necessary, leading subsequently to the risk of hypoglycemia and thus an excessive feeling of hunger. Increased energy intake and obesity.
2. Excess insulin secretion, aggravated by insulin resistance, represents an effort for the pancreas with the risk, over time, to arrive at a deficit of insulin-dependent diabetes type 2 insulin production
3. Hyperinsulinemia is also associated with reduced lipolysis and increased lipogenesis obesity and hyperlipoproteinemia
4. Fat accumulation, especially in the abdominal region, is associated with chronic inflammation and insulin resistance by type 2 diabetes tissues and metabolic syndrome In addition to these reasons, a high GI diet, typically called Western Diet, is also generally deficient in plant foods, rich in antioxidants and photo compounds with anti-inflammatory action, without which the process of chronic organic inflammation is accelerated, even in the absence of real obesity.

DETAILED DESCRIPTION:
For these reasons, in recent years the food industry has tried, not always successfully, to experiment with alternative formulations for its products, implementing a series of techniques to reduce the GI of foods, in particular those based on cereal flour. There are different methods useful to reduce the GI; in particular, the most impacting aspects of the GI of food containing carbohydrates are the sugar content, the starch content, the type of starch, the cooking method, previous processing, pre-cooking, post-cooking cooling, soaking, particle size and fiber quantity.

Increased consumption of soluble fiber is associated with reduced absorption of sugars in the intestine and therefore a reduced GI. On the contrary, most of the fibers contained in cereals and tubers are not soluble. For this reason, the direct effect of fibers on glycemic absorption is not significant. On the other hand, whole grains generally have a lower glycemic index than refined grains and this may be due to a combination of factors such as reduced digestibility, higher starch-content resistance, and the effects of other constituents of bran (such as lipids). Insoluble fibers are also attributed to a greater satiating effect.

The determination of the glycemic index can be estimated in vitro with good accuracy through an artificial digestive apparatus, or dynamic gastric model (DGM) but the gold standard remains the analysis of the glycemic response on subjects in vivo, typically volunteers. The ISO standard 26642 guidelines of 2010 represent the gold standard for the analysis of GI in humans and consists of a few simple steps that require blood sampling to determine blood sugar at the time 0, 15, 30, 45, 60, 90, and 120 min. The GI is but the average of the proportions between the sum of the 7 areas created by placing time on the abscissa (in minutes) and the ordinate blood sugar levels at each T (expressed in mmol/L or mg/dl) after consuming the test food compared to the sum of the areas created after consuming the reference food, usually glucose.

Secondly, the modulation of the intake of sugars and calories can also be managed through alternative methods. It has been seen that, for example, different stimuli related to the sense of taste can modulate the sense of hunger and consequently the calorie intake in the following hours. This is especially true with the bitter taste. Appetite modulation due to the administration of particular foods was primarily associated with particular polymorphisms of receptor genes associated particularly with a bitter taste (TAS2R) and sweet (T1R2-T1R3). At the same time, the discovery of extra-oral receptors to recognize bitterness (extra-oral TAS2R) led the researchers to test the effects of administering particular bitter foods without the potential confounding effect of oral ingestion.

Among recent studies, some researchers have shown that the effect of reducing energy intake has not been statistically significant in a group of overweight women, at least for some types of encapsulated bitterness while others have proven that an intragastric infusion of bitters significantly reduced hunger in a group of normal-weight women. Another study, in the short term, showed instead that an administration of bitters encapsulated with the base of 'Gentiana Lutea' during the morning meal can significantly reduce the energy intake of the day.

Different types of bitters can stimulate different receptors of the TAS2R family. A recent review showed that the bitters most tested and used to determine changes in hunger and energy intake were Quinine, Denatonium Benzoate, Naringin, Secoiridoid, Hops, and Gentian. Bitter compounds, in comparison to other flavors, have proved to be the most effective in influencing eating behavior. This highlights the potential preventive role of bitter flavors in the fight against epidemic obesity. However, further studies are needed to understand which bitters are most useful for this purpose, and which subcategories of the population are most effective. Artemisia Absinthium is an edible and non-toxic plant, commonly called wormwood, for which analgesic, anti-inflammatory, and antidiabetic effects are documented. The bitter extract of this plant, if properly encapsulated, could also affect appetite regulation.The purpose of the first phase of this study is to test the GI of 3 different formulations, in the form of dietary biscuits, on 12 healthy volunteer subjects in order to calculate an average GI necessary for the company that provides the product to enrich the label with a final IG and start marketing. In the second phase, the same subjects will participate in a crossover study to test the same parameters of the first phase, with the addition of an investigation on the effects on hunger with 2 formulations of biscuits different from the first 3, one containing bitter encapsulated Artemisia Absinthium base. The chemotype of Artemisia absinthium used for the extract used is thujoni-free and therefore has no documented contraindication.

ELIGIBILITY:
Inclusion Criteria:

* Absence of allergies or intolerances to tested foods
* Absence of drugs that affect glucose metabolism. Stable doses of oral contraceptives, acetylsalicylic acid, thyroxine, mineral supplements, medications for hypertension or osteoporosis are accepted.

Criteria for exclusion:

* diagnosis or history of diabetes or reduced glucose tolerance.
* surgery or severe and acute illness in the last 3 months
* use of steroids, protease inhibitors or antipsychotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | Change from fasting glucose at time 15, 30, 45, 60, 90, 120, (180) minutes
  Variation of glucose in time for each day after the ingestion of a certain food
COEQ (Control of Eating Questionnaire) | Differences between VAS scores before food ingestion (h 9:00), before lunch (h: 13:00), and before dinner (h: 20:00)
  Variation of 20-item COEQ questionnaire 100mm VAS scales for each day after the ingestion of a certain food. Hunger, satiety, quality of life, and food craving were assessed through a 100 mm VAS-scale
Ghrelin | Change from fasting ghrelin at time 15, 30, 45, 60, 90, 120, (180)
  Variation of blood acylated and des-acylated ghrelin in time for each day after the ingestion of a certain food
GLP-1 | Change from fasting GLP-1 at time 15, 30, 45, 60, 90, 120, (180)
  Variation of blood GLP-1 in time for each day after the ingestion of a certain food

SECONDARY OUTCOMES:
Insulin | Change from fasting Insulin at time 15, 30, 45, 60, 90, 120, (180)
  Variation of blood Insulin in time for each day after the ingestion of a certain food
C-Peptide | Change from fasting C-Peptide at time 15, 30, 45, 60, 90, 120, (180)
  Variation of blood C-Peptide in time for each day after the ingestion of a certain food
Leptin | At fasting for each of the 7 days
  Assessment of fasting leptin in each day
Glycated Hemoglobin (Hb1ac) | At fasting for each of the 7 days
  Assessment of fasting Hb1ac in each day
Customer preference and satisfaction | After the ingestion for each of the 5 days with biscuits
  Assessment of subject personal taste and preferences after the ingestion of the biscuits recipes. Questions are regarding taste, smell, consistency and knowledge about functional foods

OTHER OUTCOMES:
Weight | At fasting for each of the 7 days
  Assessment of weight in each day as a potential confounding factor during statistical analyses
Body circumferences | At fasting for each of the 7 days
  Assessment of body circumferences (waist and hip) in each day as potential confounding factors during statistical analyses

CONTACTS AND LOCATIONS:
Locations (1):
- : Italy Pediatric Endocrine Service of AOU Maggiore della Carità of Novara; SCDU of Pediatrics, Department of Health Sciences, University of Eastern Piedmont, Novara, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD will be available

REFERENCES:
- [Background] Kaur B, Ranawana V, Henry J. The Glycemic Index of Rice and Rice Products: A Review, and Table of GI Values. Crit Rev Food Sci Nutr. 2016;56(2):215-36. doi: 10.1080/10408398.2012.717976. PMID 25590950
- [Background] Ludwig DS. The glycemic index: physiological mechanisms relating to obesity, diabetes, and cardiovascular disease. JAMA. 2002 May 8;287(18):2414-23. doi: 10.1001/jama.287.18.2414. PMID 11988062
- [Background] Englyst KN, Vinoy S, Englyst HN, Lang V. Glycaemic index of cereal products explained by their content of rapidly and slowly available glucose. Br J Nutr. 2003 Mar;89(3):329-40. doi: 10.1079/BJN2002786. PMID 12628028
- [Background] Sivakamasundari SK, Priyanga S, Moses JA, Anandharamakrishnan C. Impact of processing techniques on the glycemic index of rice. Crit Rev Food Sci Nutr. 2022;62(12):3323-3344. doi: 10.1080/10408398.2020.1865259. Epub 2021 Jan 27. PMID 33499662
- [Background] Soh NL, Brand-Miller J. The glycaemic index of potatoes: the effect of variety, cooking method and maturity. Eur J Clin Nutr. 1999 Apr;53(4):249-54. doi: 10.1038/sj.ejcn.1600713. PMID 10334648
- [Background] Loper HB, La Sala M, Dotson C, Steinle N. Taste perception, associated hormonal modulation, and nutrient intake. Nutr Rev. 2015 Feb;73(2):83-91. doi: 10.1093/nutrit/nuu009. PMID 26024495
- [Background] Chupeerach C, Tapanee P, On-Nom N, Temviriyanukul P, Chantong B, Reeder N, Adegoye GA, Tolar-Peterson T. The influence of TAS2R38 bitter taste gene polymorphisms on obesity risk in three racially diverse groups. Biomedicine (Taipei). 2021 Sep 1;11(3):43-49. doi: 10.37796/2211-8039.1175. eCollection 2021. PMID 35223410
- [Background] Wang Q, Liszt KI, Depoortere I. Extra-oral bitter taste receptors: New targets against obesity? Peptides. 2020 May;127:170284. doi: 10.1016/j.peptides.2020.170284. Epub 2020 Feb 21. PMID 32092303
- [Background] Peters HPF, Koppenol W, Schuring EAH, Gouka R, Mela DJ, Blom WAM. The effect of two weeks ingestion of a bitter tastant mixture on energy intake in overweight females. Appetite. 2016 Dec 1;107:268-273. doi: 10.1016/j.appet.2016.08.013. Epub 2016 Aug 10. PMID 27522037
- [Background] Deloose E, Janssen P, Corsetti M, Biesiekierski J, Masuy I, Rotondo A, Van Oudenhove L, Depoortere I, Tack J. Intragastric infusion of denatonium benzoate attenuates interdigestive gastric motility and hunger scores in healthy female volunteers. Am J Clin Nutr. 2017 Mar;105(3):580-588. doi: 10.3945/ajcn.116.138297. Epub 2017 Feb 1. PMID 28148502